CLINICAL TRIAL: NCT05258682
Title: Safety of Nebulized Combination Therapy BromAc® in COVID-19 Respiratory Disease: a Phase 1 Study
Brief Title: Safety of Nebulized Combination Therapy BromAc® in COVID-19 Respiratory Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mucpharm Pty Ltd (Industry)
Collaborators: St George Hospital, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUC-COV-003
Record Dates: First submitted 2022-02-22; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pneumonia; COVID-19; Ventilator Associated Pneumonia; COVID-19 Acute Respiratory Distress Syndrome
Keywords: mucolytic; COVID-19; COVID-19 pneumonia; Ventilator associated pneumonia; Secondary bacterial infections
MeSH Terms: conditions — COVID-19; Pneumonia, Ventilator-Associated | interventions — Bromelains; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BromAc (Experimental): BromAc (Bromelain and Acetylcysteine combination) will be administered three times (3x) per day for five (5) days in a dose escalation format via inhalation using an approved vibrating mesh nebuliser (Aerogen Pro). Dose escalation concentration levels are BromAc 125ug/20mg/ml, 250ug/20mg/ml, 375ug/20mg/ml. All levels will receive 5ml of BromAc.
  Interventions: Drug: Bromelains; Drug: Acetylcysteine

INTERVENTIONS:
Drug: Bromelains — Bromelain combined with Acetylcysteine (BromAc), administered simultaneously.
  Other Names: Bromelain
Drug: Acetylcysteine — Bromelain combined with Acetylcysteine (BromAc), administered simultaneously.
  Other Names: N-Acetylcysteine

SUMMARY:
COVID-19 has multiple facets including cytokine storm, thromboembolism and gelatinous secretions. It is known that oxygen exchange is the main problem in patients with COVID-19 and hypoxia is one of the most serious, in which patients succumb to acute respiratory distress syndrome (ARDS). In other severe respiratory disease such as ventilator associated pneumonia (VAP), formation of biofilm in the endotracheal tube causes infection to spread to the lungs, resulting in respiratory decline and high mortality. The development of gelatinous sputum plugs correlates with negative outcome. Both groups of patients still have limited therapy options. BromAc is a potent mucolytic, biofilm degrader, cleaves the glycoproteins of the SARS-CoV-2 virus (antiviral), and down regulates cytokines and chemokine in COVID-19 sputum. The investigators seek to examine the safety and attempt to gain preliminary efficacy of nebulised BromAc in moderate to severe COVID-19 and other mucus producing, severe, respiratory diseases.

DETAILED DESCRIPTION:
It is well known that oxygen exchange is a major problem in patients with COVID-19 and hypoxia is one of the most serious effects, where patients succumb from acute respiratory distress syndrome (ARDS). The development of mucinous sputum plugs in individuals infected with SARS-CoV-2 is variable in the early stages of the disease. In addition, 30-40% of patients who are in hospital have expectoration production, and in a recent study on pulmonary pathology in patients with COVID-19, subsequent tests revealed markedly increased levels of MUC1 and MUC5AC in sputum and tracheal aspirates.

Currently, there are few therapeutic agents of limited efficacy to treat or avoid the complications of COVID-19 and none directed against airway mucus. An Australian pharmaceutical company has developed BromAc for the palliative treatment of highly mucinous tumors of the appendix and lung. This drug is composed of bromelain and acetylcysteine. During pre-clinical development, the sponsor found that BromAc® rapidly dissolved and removed tumour mucin, making it a potent mucolytic. BromAc® in combination have the ability, as shown in pre-clinical studies, to remove the mucin protective framework expressed by cancer including MUC1, MUC2, MUC4, MUC5AC and MUC16. The sponsor has shown the mechanism of action of BromAc - to break peptide and glycosidic linkages and disulphide bonds in tumour produced and respiratory mucin.

In an in vitro study by the sponsor with Vero and CALU-3 cells infected by SARS-CoV-2 (MOI 1 to -4) and treated with BromAc, it was found that the drug was able to reduce the virus's ability to infect cells, demonstrating an antiviral potential for SARS-CoV-2, with 99.99% reduction in viral infectivity at low concentrations. In addition to the anti-viral effect, BromAc is a potent mucolytic. In laboratory studies, BromAc (125ug or 250ug/ml plus 20mg/ml Acetylcysteine) resulted in complete dissolution of severe COVID-19 sputum after a single application within 30 minutes. BromAc significantly down-regulated cytokines and chemokines in comparison to Acetylcysteine alone or control, specifically those important to COVID-19 cytokine storm CCL2, CCL3, IL-6, CXCL10. In vivo safety models in two species have received nebulised and intranasal BromAc up to 500ug/20mg/ml three times daily for five days, with no evidence of respiratory or systemic toxicity clinically or on histology.

This project will evaluate the mucolytic and anti-inflammatory effect of BromAc in patients with moderate to severe COVID-19 that are not on mechanical ventilation. The investigators believe that BromAc may have a role clinically in removing the proteinaceous material from the bronchi and alveoli allowing improved ventilation, gas exchange and transfer and aim to study whether this is a potential treatment for these patients.

This therapy if safe may reduce the need for ventilation or improve the outcome of ventilation (reduced pressure, faster time to extubation, reduced secondary lung injury, reduced deaths), which will be assessed in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years to 75 years old
* Admitted to hospital for management of COVID-19 with moderate or severe disease
* Positive testing by virologic test (i.e. SARS-CoV-2 based qRT-PCR)
* Clinical signs suggestive of moderate or severe disease such as oxygen saturation (SpO2) less than 93% on room air or where the participant requires oxygen support such as nasal cannulas, mask, non-rebreather mask, high flow nasal cannulas

Exclusion Criteria:

* Patients that have critical disease and are mechanically ventilated
* Undergoing other airway administered mucolytic therapy for e.g. dornase alfa within 24 hours, or are enrolled in another clinical trial for COVID-19
* Have known allergy, anaphylaxis or intolerance to pineapples, papain, bromeliads, sulphur, eggs or Acetylcysteine or any other serious allergy or intolerance to fruits or food products or any other serious allergy or allergen triggered asthma, such as dust or pollen
* Have other serious comorbidities where inclusion in the trial will subject the participant to a higher risk of adverse events, including participants with asthma (existing severe lung disease such as COPD, bronchiectasis and cystic fibrosis are not exclusion criteria)
* Pregnant women are excluded from this study because BromAc has unknown but a potential risk for adverse events in nursing infants secondary to treatment of the mother
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Are unable to give fully informed and educated consent or are unable to comply with the standard follow up procedures of a clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the treatment-emergent adverse events (AEs) of BromAc therapy following nebulised delivery | Following each nebulisation on days 1 to 5 and during follow up on days 6-15, 21, 28 and 60
  The safety and tolerability of BromAc will be assessed by characterising the symptoms or side effects of treatment (treatment-emergent adverse events) by the Common Toxicity Criteria for Adverse Events (CTCAE) v4.0

SECONDARY OUTCOMES:
Proportion of participants that proceed to invasive ventilation for deterioration of COVID-19 (need for mechanical ventilation) | Daily for 60 days
  To assess the proportion of patients following commencement of BromAc that proceed to mechanical ventilation for COVID-19
World Health Organisation (WHO) modified ordinal scale clinical score | Daily for 28 days
  Determine the clinical score by improvement or deterioration based on World Health Organisation Modified Ordinal Scale for COVID-19 over 28-days
Improvement or deterioration in oxygenation | Daily for up to 14 days
  Assess the improvement or deterioration in percentage of oxygen saturation (SpO2) whilst hospitalised vs the fraction of inspired oxygen (SpO2/FiO2 ratio)
All-cause mortality | Daily for 28 days
  Determine the all-cause mortality of patients enrolled over 28 days
Dose related toxicities | Following each nebulisation on days 1 to 5 and during follow up on days 6-15, 21, 28 and 60
  Determine the tolerated dose of BromAc within the therapeutic range for COVID-19 sputum mucolysis delivered by nebuliser
Treatment-emergent serious adverse events (SAEs) | Following each nebulisation on days 1 to 5 and during follow up on days 6-15, 21, 28 and 60
  Assess the proportion of participants with treatment-emergent serious adverse events (SAEs) by Common Toxicity Criteria for Adverse Events (CTCAE) v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Frank MP van Haren, MD, PhD, Principal Investigator — St George Hospital, Director of Intensive Care

IPD SHARING:
Plan to Share IPD: No